CLINICAL TRIAL: NCT06651697
Title: BladdEr Full OR Empty for Pelvic Radiation Therapy
Acronym: BEFORE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tyler Seibert, Radiation Oncologist, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 811100
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Neoplasm
Keywords: malignancy of the pelvis; bladder; radiation therapy
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full bladder (Active Comparator): Full bladder protocol for participants undergoing radiation therapy to pelvis for common malignancies.
  Interventions: Radiation: Radiation therapy
- Empty bladder (Experimental): Empty bladder protocol for participants undergoing radiation therapy to pelvis for common malignancies.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy with full bladder or empty bladder protocols

SUMMARY:
The present study evaluates empty and full bladder protocols for radiation therapy of genitourinary (GU), gynecological (Gyn), and gastrointestinal (GI) malignancies of the pelvis.

DETAILED DESCRIPTION:
Pelvic radiation therapy plays a key role in the treatment of common genitourinary (GU), gynecological (Gyn), and gastrointestinal (GI) malignancies of the pelvis. Prior to starting a course of radiation therapy, patients undergo a CT simulation that allows for computer-based optimization of radiation dose delivery to target while simultaneously minimizing dose to surrounding normal tissues, such as the bladder and rectum. Commonly, physicians instruct patients undergoing pelvic radiation therapy to present with a reproducibly full bladder for the simulation and for each subsequent treatment session with the hope that increased distance between normal tissues (anterior bladder wall and bowel) and treatment target will limit toxicity. However, treating with a full bladder can result in wide variations in bladder volume. Often patients are unable to reproduce the bladder distention achieved at simulation, especially as typical urinary symptoms related to radiation develop during treatment. As the initial CT simulation is used to calculate dose distribution, bladder volume changes can affect radiation dose distribution to the bladder itself as well as adjacent pelvic organs. Given the challenges and uncertainties of treating with a full bladder, there has been increasing interest in bladder empty protocols. Retrospective, non-randomized, single-institution studies demonstrate that bladder empty protocols reduced absolute variation in bladder volume during treatment, had minimal impact on treatment related toxicity, and had non-inferior biochemical progression free survival, GI toxicities, and GU toxicities. However, prospective data is very limited. The present study plans to fill this knowledge gap by randomizing study participants to empty and full bladder protocols for simulation and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Persons, aged at least 18 years
* Deemed eligible to undergo curative intent radiation therapy for primary GU, GI, or Gyn malignancy of the pelvis.
* For participants able to become pregnant: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation
* For participants able to cause a pregnancy: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

* Pregnancy
* Tumor invading the bladder, as judged by the enrolling physician based on available clinical information
* Contraindications to radiotherapy, including Crohn's disease and active connective tissue disorders such as scleroderma or uncontrolled lupus
* Prior radiation therapy to an area requiring treatment in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 3 months post radiation
  Acute any attribution GU and/or GI grade ≥2 toxicity. This will be defined as the percentage of patients with CTCAE version 5.0 GU and/or GI grade ≥2 toxicity within 3 months post radiation therapy. This will be defined as a co-primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Seibert, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available